CLINICAL TRIAL: NCT00345007
Title: Assessment of Recovery of Macula Function After Successful Scleral Buckling Surgery for Rhegmatogenous Retinal Detachment
Brief Title: Macular Function After Scleral Buckle
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R414/09/2005
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2005-05

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Retinal detachment; Macular function; Multifocal electrophysiology
MeSH Terms: conditions — Retinal Detachment | interventions — Scleral Buckling

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Scleral buckling

SUMMARY:
Assess recovery of macula function after successful scleral buckling surgery for rhegmatogenous retinal detachment by using the multifocal ERG in the postoperative period i.e. recovery of functional integrity 2. Assess the relationship between the neurosensory retina and the retinal pigment epithelium/choriocapillaris after scleral buckling i.e. recovery of structural integrity 3. Assess if there is a difference between macula function postoperatively, in eyes with retinal detachments involving the macula and those that do not.

DETAILED DESCRIPTION:
Patients with acute rhegmatogenous retinal detachments managed by scleral buckling surgery will be recruited into 3 groups. (Please see attached appendix A)

We define the area of the macula as the area within the temporal vascular arcades with the horizontal radius defined between the optic disc and the foveal centre.

Group A: Macula not detached Group B: Macula partially detached i.e. detachment stops within the macula Group C: Macula is totally detached

After scleral buckling surgery for the retinal detachment, the patients will be examined at Day 1, week 1, month1, 3 and 6. During these visits, they will be examined clinically, as well as undergo tests - refraction, colour vision (D-15) & contrast sensitivity testing, OCT and multifocal ERG. (Please see attaced visit schedule).

ELIGIBILITY:
Inclusion Criteria:

* Acute rhegmatogenous retinal detachment undergoing scleral buckling surgery

Exclusion Criteria:

* Only eye patients
* Patients who undergo surgery which require use of intravitreal gases
* Patients who will not be able to cooperate for the mfERG and OCT testing
* Patients with macula hole detachments
* Fellow eye with poor vision resulting in inability to fixate for the mfERG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2005-06; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yen Lee, FRCSEd, Principal Investigator — Singapore National Eye Centre; Chong-Lye Ang, FRCOphth, Study Chair — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore